CLINICAL TRIAL: NCT04110405
Title: Scaling-Up Stepped Care for Women's Mental Health in Primary Care in an LMIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Prisma Research Center (Unknown); University of Utah (Other); New York University (Other)
Responsible Party: Principal Investigator, Stevan Weine, Professor of Psychiatry, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0745
Record Dates: First submitted 2019-09-18; First posted 2019-10-01 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped Care (Experimental): To assess the effectiveness of the stepped care model with 420 women who have depression and potential co-occurring anxiety, recruited from 12 primary care clinics in Tajikistan.
  Interventions: Behavioral: Stepped Care
- Standard of Care plus Healthy Lifestyle (Active Comparator): To compare standard of care plus healthy lifestyle materials with 210 women recruited from 6 primary care clinics in Tajikistan.
  Interventions: Behavioral: Standard of Care plus Healthy Lifestyle

INTERVENTIONS:
Behavioral: Stepped Care — This stepped care model involves three steps. Step 1 is a peer and nurse co-led 8-session group based upon BRIDGES. Step 2 is peer or nurse led 6-session individual meetings based upon Interpersonal Psychotherapy. Step 3 is primary care physician led medication treatment with Amitriptyline.
  Arms: Stepped Care
Behavioral: Standard of Care plus Healthy Lifestyle — Standard outpatient care supplemented with literature on healthy lifestyles will serve as an enhanced control condition. In each clinic, non-specialty mental health care is available in the form of counseling from doctors or nurses along with psychiatric medication management. Given the difficulties faced by women in Tajikistan, ethical responsibility compels us to enhance the control condition by having nurses distribute written materials on healthy eating, physical fitness, and personal hygiene, at a reading level which will be widely accessible.
  Arms: Standard of Care plus Healthy Lifestyle

SUMMARY:
This study examines: 1) short-term and longitudinal impacts of stepped care on women with depression and the possible roles of mediators and moderators; 2) clinic- (readiness to adopt an innovation, leadership support and climate) and provider-level (preparedness, motivation and fidelity) factors that may affect stepped care implementation; and 3) the differential impact of two implementation approaches (a clinic implementation teams versus implementation training by the research team). It utilizes Curran's hybrid effectiveness implementation design, mixed methods, and a longitudinal design with assessments at pre, 3 months, 6 months, and 12 months. A total of 18 primary care clinics, set in both rural and urban communities in Tajikistan, will be involved, with 12 delivering the intervention and 6 acting as controls. 8 providers (3 nurses, 3 peers, and 2 doctors) will be recruited at each of the 12 intervention clinics for a total of 96 providers; 35 women with depression will be recruited from each clinic for a total of 630 women.

DETAILED DESCRIPTION:
This research will advance mental healthcare task sharing in effectiveness and implementation testing of a stepped care model for LMICs. It uses nurses and mental health peers to treat depression and potential co-occurring anxiety among women in primary care. The study addresses Grand Challenges in Global Mental Health Goal C to foster integration of mental health into primary care and NIMH Strategic Aim 3 by developing new and better interventions that incorporate the diverse needs and circumstances of people with mental illness. It utilizes Curran's hybrid effectiveness implementation design. To improve implementation, it examines the impact of clinic implementation teams in readying the clinic and service providers. Additionally, it explores how RDoC neuroscience contributes to implementation science through enhancing the evaluation and targeting of stepped care. This study will enable new collaborative research activities, in tandem with network building, mentorship and training, and dissemination of findings, which will further build the LMIC capacity for implementation science research and development of evidence-based medicine by strengthening Tajikistan's individual and institutional research capabilities.

Globally, young women bear a disproportionate burden of common mental disorders, and especially including depression and potentially co-occurring anxiety. With current care models, this burden cannot be lifted without finding ways to deliver mental health prevention and treatment services and illness self-management to women in primary care. Our previous research in Tajikistan has demonstrated that women are exposed to serious risks for mental illness, and how peers and primary care nurses have played major but largely informal roles in helping women with mental health problems. Therefore, the investigators developed and tested for feasibility a stepped care model which showed very strong treatment effects. This stepped care model involves three steps. Step 1 is a peer and nurse co-led 8-session group based upon BRIDGES. Step 2 is peer or nurse led 6-session individual meetings based upon Interpersonal Psychotherapy. Step 3 is primary care physician led medication treatment with Amitriptyline.

This project will scale-up the intervention in multiple polyclinics, so as to examine its effectiveness (Aim 2) and to compare two implementation strategies (Aim 3). This presents a remarkable opportunity to advance both services and science of mental health in Tajikistan.

Aim 1. To assess the effectiveness of the stepped care model with 420 women who have depression and potential co-occurring anxiety, recruited from 12 primary care clinics in Tajikistan, compared with standard of care plus provision of healthy lifestyle materials, with another 210 women recruited from 6 primary care clinics, including assessing mediators and moderators (e.g. executive control efficiency, trauma exposure).

Aim 2. To assess whether a clinic implementation team moderates women's reduction in depression post-intervention, as well as clinic-level (leadership support and degree of implementation) and provider-level (motivation and fidelity) moderators.

Aim 3. To establish a national mental health research network that focuses on improving the standard of mental health care and access to services by building mental health implementation research capacity.

ELIGIBILITY:
Inclusion Criteria:

* female Tajik citizen between 18 and 45 years old
* score >16 on the HAM-D
* no current or past substance use
* willing to participate in the intervention and research procedures
* able to give written informed consent.

Exclusion Criteria:

* women who are older or younger than 18 - 45 years
* women who do not score >16 on the HAM-D

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Self-representation of gender identity
Enrollment: 630 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
change in Hamilton Depression Rating Scale | baseline, 3 months, 6 months, and 12 months
  The Hamilton Depression Rating Scale (HAM-D) is a way of determining a patient's level of depression before, during, and after treatment. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2. Score of 0-7 = normal; 8-13 = mild depression; 14-18 = moderate depression; 19-22 = severe depression, +23 = very severe depression.
change in Texas Christian University (TCU) Organizational Readiness for Change | baseline, 3 months, 6 months, and 12 months
  Motivational factors include program needs, training needs, and pressures for change, while program resources are evaluated in regard to office facilities, staffing, training, equipment, and the Internet. Organizational dynamics include scales on staff attributes and climate.
  Numbers for each item indicate its location in the administration version, in which response categories are 1=Strongly Disagree to 5=Strongly Agree; ® designates items with reflected scoring. Scores for each scale are obtained by summing responses to its set of items (after reversing scores on reflected items by subtracting the item response from "6"), dividing the sum by number of items included (yielding an average) and multiplying by 10 in order to rescale final scores so they range from 10 to 50 (e.g., an average response of 2.6 for a scale becomes a score of "26").

SECONDARY OUTCOMES:
change in Hamilton Anxiety Rating Scale | baseline, 3 months, 6 months, and 12 months
  The Hamilton Anxiety Rating Scale (HAM-A) measures the severity of anxiety symptoms. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity, and 25-30 moderate to severe.
change in PTSD Checklist for DSM- 5 | baseline, 3 months, 6 months, and 12 months
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including monitoring symptom change during and after treatment, screening individuals for PTSD, making a provisional PTSD diagnosis.Respondents are asked to rate how bothered they have been by each of 20 items in the past month on a 5- point Likert scale ranging from 0 not at all, 1 a little bit, 2 moderately, 3 quite a bit, 4 extremely. Items are summed to provide a total severity score (range = 0-80).Summing all 20 items and using cut-point score of 33 appears to be reasonable based upon current psychometric work.
change in Evidence Based Practice Attitude Scale | baseline, 3 months, 6 months, and 12 months
  This tool (EBPAS) examines attitudes toward evidence-based practice among social service providers. The tool includes 15 questions regarding clinician and case manager willingness to adopt evidence-based practices given the appeal of evidence-based practice, system, organization, or supervisor requirements for evidence-based practices. The four scales are labeled as "Requirements scale" (3 items), "Appeal scale" (4 items), "Openness scale" (4 items), "Divergence scale" (4 items). A higher score indicates "more" of the scale name, except for Divergence
# Stepped Care interventions initiated and completed | baseline, 3 months, 6 months, and 12 months
  Measure the number of stepped care interventions that were initiated and those that were completed.

CONTACTS AND LOCATIONS:
Locations (20):
- Tajikistan (20):
  - City Health Center #4, Dushanbe
  - City Health Center #5, Dushanbe
  - Dushanbe City Health Center #12, Dushanbe
  - Dushanbe City Health Center #13, Dushanbe
  - Dushanbe City Health Center #15, Dushanbe
  - Dushanbe City Health Center #1, Dushanbe
  - Dushanbe City Health Center #2, Dushanbe
  - Dushanbe City Health Center #6, Dushanbe
  - Guliston District Health Center, Guliston
  - Gafurov District Health Center, Khujand
  - Kayrokum District Health Center #7, Khujand
  - Khujand City Health Center #1, Khujand
  - Khujand City Health Center #2, Khujand
  - Khujand City Health Center #3, Khujand
  - Khujand City Health Center #4, Khujand
  - Khujand City Health Center #5, Khujand
  - Khujand City Health Center #6, Khujand
  - Rudaki District Health Center, Rŭdakí
  - Shahrinav District Health Center, Shahrinav
  - Varzob District Health Center, Varzob

IPD SHARING:
Plan to Share IPD: No